CLINICAL TRIAL: NCT00832091
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Response Study of the Safety and Efficacy of Thymosin Beta 4 in the Treatment of Patients With Venous Stasis Ulcers
Brief Title: Study of Thymosin Beta 4 in Patients With Venous Stasis Ulcers
Acronym: SSVS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RegeneRx Biopharmaceuticals, Inc. (Industry)
Collaborators: sigma-tau i.f.r. S.p.A. (Industry)
Responsible Party: Dr Giorgio Guarnera, Istituto Dermopatico dell'Immacolata (IDI), Rome, ITaly
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SSVS
Record Dates: First submitted 2009-01-28; First posted 2009-01-29 (Estimated); Results first posted 2010-03-24 (Estimated); Last update posted 2010-03-30 (Estimated); Status verified 2010-03

CONDITIONS: Venous Stasis Ulcers
Keywords: Venous Stasis Ulcers; venous insufficiency; leg ulcers; Thymosin Beta 4; Laminin-5
MeSH Terms: conditions — Varicose Ulcer; Venous Insufficiency; Leg Ulcer | interventions — thymosin beta(4); Gels

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): There are 3 groups of patients with venous stasis (VS) ulcers. Each group included 18 patients receiving active drug and 6 receiving placebo. There were 3 concentrations used for topical administration to the active drug groups: 0.01% weight/weight (w/w), 0.03% w/w, and 0.1% w/w thymosin beta 4 gel applied once daily for up to 84 days
  Interventions: Drug: Thymosin Beta 4
- 2 (Placebo Comparator): There were 3 groups of patients with venous stasis (VS) ulcers. Each group included 18 patients receiving active drug and 6 receiving placebo. There was one concentration of placebo gel for topical administration to the placebo group. The concentration was 0.0% weight/weight (w/w) thymosin beta 4 gel applied once daily for up to 84 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Thymosin Beta 4 — There were 3 groups of patients with venous stasis (VS) ulcers. Each group included 18 patients receiving active drug and 6 receiving placebo. There were three concentrations of gel used for topical administration to the active groups: 0.01% weight/weight (w/w), 0.03% w/w, and 0.1% w/w thymosin beta 4 gel applied once daily for up to 84 days
  Other Names: Tβ4; RGN-137 (topical gel)
  Arms: 1
Drug: Placebo — There were 3 groups of patients with venous stasis (VS) ulcers. Each group included 18 patients receiving active drug and 6 receiving placebo. There was one concentration of placebo gel for topical administration to the placebo group. The concentration was 0.0% weight/weight (w/w) thymosin beta 4 gel applied once daily for up to 84 days
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and effectiveness of Thymosin Beta 4 administered topically in patients with Venous Stasis ulcers

DETAILED DESCRIPTION:
The purpose of this double-blind, placebo-controlled, dose-response study is to evaluate the safety, tolerability and effectiveness of Thymosin Beta 4 (Tβ4), administered topically, in patients with Venous Stasis (VS) ulcers. VS ulcers develop on the ankle or lower leg in patients with chronic vascular disease. In these patients, blood flow in the lower extremities is impaired, leading to edema (swelling) and mild redness and scaling of the skin that gradually progress to ulceration. Tβ4 is a synthetically-produced copy of a naturally occurring 43 amino acid peptide that has wound healing and anti-inflammatory properties and can up-regulate the expression of laminin-5.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent Form signed by the patient
* Male or female, between 18 and 79 years of age
* At least one venous leg ulceration stable for at least 6 weeks before enrollment
* Surface area between 3 and 30 cm2

Exclusion Criteria:

* Have clinical evidence of active infection on the index ulcer
* Use of any experimental drug, or participation in any clinical study, within the 60 days before enrollment
* Use of systemic or topical steroidal therapy, immunotherapy, or cytotoxic chemotherapy within the 60 days before enrollment
* History of adverse reaction to any ingredients of the study medication
* Clinically significant neurological, cardiovascular, respiratory, hepatic, renal, metabolic and dermatologic disease other than venous ulcers
* Current or former malignancy
* Arterial disorder resulting in ulcerated ulcers
* Diabetes mellitus
* Pregnant or lactating (breastfeeding) women. A serum pregnancy test will be performed at screening for female patients of childbearing potential

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2006-07; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Guarnera, MD, Principal Investigator — Istituto Dermopatico Dell'Immacolata, Rome , Italy
Locations (8):
- Italy (5):
  - Chirurgia Vascolare, Bologna
  - Università degli Studi di Napoli - Federico II, Naples
  - Azienda Ospedaliera di Padova, Padua
  - Unità Operativa di Angiologia Azienda Ospedaliera di Padova, Padua
  - Istituto Dermopatico dell'Immacolata (IDI), Rome
- Poland (3):
  - Klinika Chirurgii Naczyń i Angiologii, Lublin
  - Klinika Chirurgii Ogólnej i Naczyniowej,, Szczecin
  - Oddział Angiologiczny, Wroclaw

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started in 2006 and ended in 2009 using 8 sites: University Medical Center Clinics
Pre-assignment Details: Prior to randomization, patients need to meet specific inclusion and exclusion criteria. There was no wash-out or run-in periods
Groups:
- Placebo: 0.00% Thymosin Beta 4 (Tβ4), weight/weight (w/w)
- Thymosin Beta 4 (Tβ4) at 3 Doses: 0.01% Tβ4 weight by weight (w/w), 0.03% Tβ4 w/w, 0.1% Tβ4 w/w
Period: Overall Study
Arm/Group | Placebo | Thymosin Beta 4 (Tβ4) at 3 Doses
Started | 17 | 55
Completed | 12 | 53
Not Completed | 5 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Prohibited Medication | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Thymosin Beta 4 (Tβ4) at 3 Doses | Total
Number analyzed (Participants) | 17 | 55 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 39 | 48
  >=65 years | 8 | 16 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 28 | 40
  Male | 5 | 27 | 32
Region of Enrollment [Number; unit: participants]
  Poland | 6 | 38 | 44
  Italy | 11 | 17 | 28

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Thymosin Beta 4 (Tβ4) Applied to Patients With Venous Stasis (VS) Ulcers for up to 84 Days
Description: All Treatment-Emergent (TE) Serious Adverse Events (SAEs) and Adverse Events (AEs) by treatment with Tβ4 gel at the combined 3 doses in the safety population with Venous Stasis (VS) ulcers for up to 84 days. TEAE is defined as a side effect that begins or that worsens in severity after the application of at least one dose of Tβ4 gel on the venous stasis ulcer. A pre-existing condition is not considered an AE, but if it worsens during the study, then it may be considered an AE
Time Frame: Up to 84 days
Population: Analysis per protocol, ITT, using LOCF
Measure: Number; unit: SAEs and AEs
Arm/Group | Placebo | Thymosin Beta 4 (Tβ4) at 3 Doses
Number analyzed (Participants) | 17 | 55
SAEs and AEs | 24 | 104

2. Secondary Outcome: Wound Healing (Wound Closure Without Drainage) by Applying Tβ4 Gel Once Daily for up to 84 Days to Patients With Venous Stasis (VS) Ulcers
Description: Wound healing effectiveness of Tβ4 gel applied once daily for up to 84 days to patients expressed as the number of patients whose wound had closed without drainage at the end of the study, Day 84
Time Frame: Up to 84 days
Population: Analysis per protocol, Intent-to-treat (ITT), using Last Observation Carried Forward (LOCF)
Measure: Number; unit: Participants
Arm/Group | Placebo | Thymosin Beta 4 (Tβ4) at 3 Doses
Number analyzed (Participants) | 17 | 55
Participants | 4 | 12

ADVERSE EVENTS:
Time Frame: 99 days
Arm/Group | Placebo | Thymosin Beta 4 (Tβ4) at 3 Doses
Serious Adverse Events (participants affected / at risk) | 1/17 | 3/55
Other Adverse Events (participants affected / at risk) | 11/17 | 35/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=17) | Thymosin Beta 4 (Tβ4) at 3 Doses (N=55)
Connective tissue, inflammation (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) — SAE not related to TB4
Increased Transamines (Investigations) | 1 (1) | 0 (0) — SAE not related to TB4
Lymphangitis (Infections and infestations) | 1 (2) | 0 (0) — SAE not related to TB4
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (4) — SAE not related to TB4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=17) | Thymosin Beta 4 (Tβ4) at 3 Doses (N=55)
Mycobacterium ulcerans infection (Infections and infestations) | 0 (0) | 1 (1)
Red blood cell sedimentation rate increased (Investigations) | 0 (0) | 6 (6)
alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
bilirubin conjugated increased (Investigations) | 0 (0) | 1 (1)
blood calcium decreased (Investigations) | 0 (0) | 1 (1)
blood creatinine phosphokinase increased (Investigations) | 1 (1) | 3 (3)
blood potassium increased (Investigations) | 1 (1) | 0 (0)
body temperature increased (Investigations) | 1 (1) | 0 (0)
bronchitis acute (Infections and infestations) | 0 (0) | 2 (3)
cystitis (Infections and infestations) | 1 (1) | 0 (0)
gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
genitourinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
helicobacter gastritis (Infections and infestations) | 0 (0) | 1 (1)
in urine protein/creatinine ratio increased (Investigations) | 0 (0) | 1 (1)
influenza (Infections and infestations) | 1 (1) | 0 (0)
inviral infection (Infections and infestations) | 0 (0) | 1 (2)
nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2)
platelet count increased (Investigations) | 1 (1) | 0 (0)
pulpitis dental (Infections and infestations) | 0 (0) | 1 (1)
red blood cell count increased (Investigations) | 0 (0) | 1 (1)
upper respiratory infection (Infections and infestations) | 0 (0) | 3 (3)
urinary sediment present (Investigations) | 0 (0) | 1 (1)
urinary tract infection (Infections and infestations) | 0 (0) | 3 (3)
white blood cell count decreased (Investigations) | 0 (0) | 1 (1)
white blood cell increased (Investigations) | 0 (0) | 2 (2)
white blood cell urine positive (Investigations) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)
erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (5)
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — AE not related to TB4
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — AE nnot related to TB4
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — AE not related to TB4
rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — AE not related to TB4
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — AE nt related to TB4
venous ulcer pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Inflammation (General disorders) | 1 (1) | 4 (5)
face edema (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 1 (1) | 1 (2) — AE not related to TB4
edema peripheral (General disorders) | 1 (1) | 0 (0)
pyrexia (General disorders) | 0 (0) | 1 (1)
Secretion Discharge (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Pain in extremities (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — AE not related to TB4
Varicose ulceration (Vascular disorders) | 1 (1) | 2 (4)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 1 (2)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Gingivitis (Gastrointestinal disorders) | 1 (1) | 0 (0) — AE not related to TB4
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypercholesteroloemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1) — AE not associated with TB4
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Renal Failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 1 (1) — AE unrelated to TB4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
RegeneRx/Sigma-Tau agreements may vary with individual investigators, but will not prohibit any investigator from publishing. RegeneRx/Sigma-Tau support the publication of results from all centers of a multi-center trial but requests that reports based on a single-site data not precede the primary publication of the entire clinical trial.